CLINICAL TRIAL: NCT06360289
Title: Observational Study of Neurofilament Light Chain (NfL) Levels in Asymptomatic Carriers of the TTR Gene Variants and Patients With hATTR Amyloidosis With Polyneuropathy, Including Patients Who Undergo Treatment Change - NeuroFeeL Study
Brief Title: Observational Study of Neurofilament Light Chain (NfL) as a Biomarker in Asymptomatic Carriers of the Transthyretin (TTR) Variants and Patients With Hereditary Transthyretin-mediated (hATTR) Amyloidosis With Polyneuropathy
Status: Recruiting | Type: Observational
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ALN-TTR-NT-003
Record Dates: First submitted 2024-04-08; First posted 2024-04-11 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Hereditary Amyloidosis, Transthyretin-Related; Asymptomatic Carrier State
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asymptomatic Carriers: Participants who are asymptomatic carriers of a pathogenic TTR variant, and not diagnosed with hATTR amyloidosis with polyneuropathy will be enrolled in this cohort.
  Interventions: Other: Standard of Care
- Participants with hATTR Amyloidosis with Polyneuropathy: Participants with a confirmed diagnosis of hATTR amyloidosis with polyneuropathy with a documented TTR variant will be enrolled in this cohort.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Standard of Care — This is an observational study. No study drug will be administered as a part of the study, participants will be treated according to the decision of the treating physician.

SUMMARY:
This is a single-center observational study evaluating the potential value of NfL as a biomarker for diagnosis, detection of disease onset, monitoring of disease progression, and treatment response in asymptomatic carriers of TTR variants and symptomatic hATTR amyloidosis patients with polyneuropathy.

DETAILED DESCRIPTION:
In this study, participants' data will be extracted from their medical records or collected based on clinical and laboratory assessments during routine visits, per the site's standard of care. Blood samples collected from the participants during routine visits will also be used for analysis. The study will be conducted in two parts: Cross-Sectional part during which a single measurement of NfL levels will be performed using blood samples collected from asymptomatic carriers, and symptomatic hATTR amyloidosis patients; Longitudinal part during which measurements of NfL levels will be performed over time using blood samples (already collected from the participants during routine visits) from asymptomatic carriers and patients with symptomatic hATTR amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

- Carrier of a documented pathogenic TTR variant confirmed with genotyping with predicted disease onset within 5 years and not diagnosed with hATTR amyloidosis with polyneuropathy

OR

Confirmed diagnosis of hATTR amyloidosis with polyneuropathy with a documented TTR variant confirmed with genotyping

- Participant is able to understand the study and does not oppose participating in the study after reviewing the content of the PIS provided.

Exclusion Criteria:

* A known condition (other than hATTR amyloidosis) that can cause nerve damage and affect NfL levels
* Estimated glomerular filtration rate (eGFR) <45 milliliters per minute per 1.73 meters squared (mL/min/1.73 m^2)
* Currently enrolled in a clinical study for any investigational agent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study will include asymptomatic carriers of TTR variants or symptomatic patients with hATTR amyloidosis with polyneuropathy who review and confirm their understanding of the Patient Information Sheet (PIS) provided and do not oppose participating in the study at Centre Hospitalier Universitaire (CHU) Le Kremlin-Bicêtre Assistance Publique-Hôpitaux de Paris (APHP).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
NfL Levels in Asymptomatic Carriers of a TTR Variant and Symptomatic hATTR Patients With Polyneuropathy at Baseline | Baseline
Change in NfL Levels Over Time in Asymptomatic Carriers of a TTR Variant and Symptomatic hATTR Patients With Polyneuropathy | Up to 24 months

SECONDARY OUTCOMES:
Correlation Between the NfL Levels and Various Biological and Clinical Activity Parameters in Asymptomatic Carriers of a TTR Variant and Symptomatic hATTR Patients With Polyneuropathy at Baseline | Baseline
Correlation Between the Change in NfL Levels and Various Biological and Clinical Activity Parameters in Asymptomatic Carriers of a TTR Variant and Symptomatic hATTR Patients With Polyneuropathy | Up to 24 months
Comparison of the Measured NfL Levels to the Normal Levels Expected to be Seen in the General Population by Using the Existing Reference Ranges and Databases | Baseline, 24 months
Time to Onset of Active Disease in Asymptomatic Carriers of TTR Variants | Up to 24 Months
Disease Progression in Symptomatic hATTR Amyloidosis Patients with Polyneuropathy | Up to 24 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire (CHU) Le Kremlin-Bicêtre Assistance Publique-Hôpitaux de Paris (APHP), Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No